CLINICAL TRIAL: NCT04068038
Title: Pediatric Acute Respiratory Distress Syndrome: a Prospective Asian Multicenter Study
Brief Title: Pediatric Acute Respiratory Distress Syndrome Asia Study
Acronym: PARDS Asia
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Guangzhou Women and Children's Medical Center (Other); Shengjing Hospital (Other); Children's Hospital of Fudan University (Other); Hong Kong Children's Hospital (Other); Sarawak General Hospital (Other); Universiti Kebangsaan Malaysia Medical Centre (Other); University of Malaya (Other); King Chulalongkorn Memorial Hospital (Other); Siriraj Hospital (Other); Ramathibodi Hospital (Other); National Children's Hospital, Vietnam (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Rumah Sakit Anak dan Bunda Harapan Kita (Unknown); Sanglah General Hospital (Other); General Hospital of North Sumatera University (Unknown); Hyogo Prefectural Kobe Children's Hospital (Other); Aga Khan University (Other); National University Hospital, Singapore (Other); Singapore Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Judith Wong Ju-Ming, Consultant Pediatric Critical Care, KK Women's and Children's Hospital
Other Study IDs: 2017/3076(2)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Distress Syndrome; Pediatric Intensive Care Unit; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — Respiratory fluid Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ventilation protocol — An evidence based ventilation protocol will be implemented at participating sites. This will include limits on peak inspiratory pressure (28cmH2O), driving pressure (16cmH2O), tidal volume (mild 8ml/kg, mod/severe 6ml/kg), positive end expiratory pressure to fraction of inspired oxygen table, permissive hypercarbia (mild allow pH 7.30, mod/severe allow pH 7.20) and permissive hypoxia (mild SpO2 92-97%, mod/severe SpO2 88-92%).

SUMMARY:
Mortality rates in children with pediatric acute respiratory distress syndrome (PARDS) are higher in Asia compared to other regions. In adults with acute respiratory distress syndrome, the only therapy that improves mortality rates is a lung protective ventilation strategy. The pediatric ventilation recommendations are extrapolated from evidence in adults, including ventilation with low tidal volume, low peak/plateau pressures and high-end expiratory pressure. A recent retrospective study of ventilation practices in Asia showed varying practices with regards to pulmonary and non-pulmonary therapies, including ventilation. This study aims to determine the prevalence and outcomes of PARDS in the Pediatric Acute and Critical Care Medicine Asian Network (PACCMAN). This study will also determine the use of pulmonary (mechanical ventilation, steroids, neuromuscular blockade, surfactant, pulmonary vasodilators, prone positioning) and non-pulmonary (nutrition, sedation, fluid management, transfusion) PARDS therapies. To achieve this aim, a prospective observational study which involves systematic screening of all pediatric intensive care unit (PICU) admissions and collection of pertinent clinical data will be conducted. Recruitment will be consecutive and follow up will continue to intensive care discharge.

DETAILED DESCRIPTION:
The overall objective of this study is to prospectively determine the epidemiology of children with PARDS and describe its management in Asia. The first specific aim is to determine the prevalence of PARDS among PICU admissions. This will be achieved by establishing a systematic manner of screening patients and including them in this study. The second specific aim is to describe the use of pulmonary and non-pulmonary therapies in PARDS. This study will utilize an established dataset to extract pertinent and analyzable clinical data.The third specific aim is to determine the outcome of patients with PARDS. These outcomes will include functional data, PICU mortality, ventilator duration and length of stay data. This is a two-part study - the first part to establish the baseline prevalence and ventilator management strategies, the second part will include the implementation of an evidence based ventilation protocol as part of routine care. The same screening process, eligibility criteria and data collection will apply throughout the two parts. We aim to obtain data for approximately 2years prior to and 2years subsequent to the implementation of the ventilator protocol.

ELIGIBILITY:
Inclusion Criteria:

* Satisfies the Pediatric Acute Lung Injury Consensus Conference (PALICC) criteria for PARDS

Exclusion Criteria:

* Premature neonates with a corrected age of less than 33 weeks and perinatal lung disease
* High flow nasal cannula

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All PICU admission will be screened daily and those who meet the PALICC criteria for PARDS will be recruited and consented (if necessary). We will include those on non-invasive ventilation and alternative modes of ventilation. However, a minimum positive end expiratory pressure of 5cmH2O is necessary for inclusion, as per PALICC. Patients with any type of cardiorespiratory comorbidity will also be included if they fulfill the PALICC criteria for special populations (cyanotic heart disease, chronic lung disease and left ventricular failure). Patients who have limitation of care (i.e. do-not-resuscitate orders) or develop brainstem death will also be included to enable calculation of prevalence.
Sampling Method: Non-Probability Sample
Enrollment: 738 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of PARDS | Through study completion
  Number of participants diagnosed with PARDS over number of intensive care admissions
Mortality | up to 60 days
  Number of PARDS participants who died over number of participants diagnosed with PARDS

SECONDARY OUTCOMES:
Ventilator free days | up to 28 days
  Number of days alive and free of mechanical ventilation
Intensive Care Unit free days | up to 28 days
  Number of days alive and discharge from the intensive care unit
Extracorporeal membrane oxygenation | up to 28 days
  Number of participants who require ECMO

OTHER OUTCOMES:
Composite mortality and ECMO | up to 60 days
  Number of PARDS participants who died or required ECMO over total number of participants diagnosed with PARDS
Sensitivity analysis | up to 60 days
  Mortality and secondary outcomes excluding limitation of care orders

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ju Ming Wong, Principal Investigator — KK Women's and Children's Hospital
Locations (19):
- China (4):
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangzhou
  - Shengjing hospital of China Medical University, Shenyang, Liaoning
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chongqing Hospital, Chongqing, Sichuan
- Hong Kong Children's Hospital, Kowloon Bay, Kowloon, Hong Kong
- Post Graduate Institute of Medical Education and Research, Chandigarh, India
- Indonesia (2):
  - Sanglah Hospital Denpasar, Denpasar, Bali
  - Harapan Kita Children and Women hospital, Jakarta
- Hyogo Prefectural Kobe Children's Hospital, Hyōgo, Kobe, Japan
- Malaysia (3):
  - Universiti Kebangsaan Malaysia Medical Centre, Bandar Tun Razak, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
  - University Malaya Medical Centre, Kuala Lumpur
- Aga Khan University Hospital, Karachi, Pakistan
- Singapore (2):
  - KK Women's and Children's Hospital, Singapore
  - National University Hospital, Singapore, Singapore
- Thailand (3):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi hospital, Bangkok
- National Hospital of Pediatrics, Đống Đa, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing will depend on ethics approval of individual sites

REFERENCES:
- [Derived] Wong JJM, Dang H, Gan CS, Phan PH, Kurosawa H, Aoki K, Lee SW, Ong JSM, Fan LJ, Tai CW, Chuah SL, Lee PC, Chor YK, Ngu L, Anantasit N, Liu C, Xu W, Wati DK, Gede SIB, Jayashree M, Liauw F, Pon KM, Huang L, Chong JY, Zhu X, Hon KLE, Leung KKY, Samransamruajkit R, Cheung YB, Lee JH; Pediatric Acute & Critical Care Medicine Asian Network (PACCMAN). Lung-Protective Ventilation for Pediatric Acute Respiratory Distress Syndrome: A Nonrandomized Controlled Trial. Crit Care Med. 2024 Oct 1;52(10):1602-1611. doi: 10.1097/CCM.0000000000006357. Epub 2024 Jun 26. PMID 38920618